CLINICAL TRIAL: NCT06507618
Title: A Randomized, Phase III Trial of Pre-Operative Window of Endocrine Therapy to Inform Radiation Therapy Decisions in Older Women With Early-Stage Breast Cancer (POWER II)
Brief Title: Pre-Operative Window of ET to Inform RT Decisions (POWER II)
Acronym: POWER II
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Shayna Showalter, MD, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR230513
Record Dates: First submitted 2024-06-20; First posted 2024-07-18 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Female
Keywords: breast cancer; endocrine therapy; radiation; letrozole; anastrozole; exemestane; tamoxifen; survey; questionnaire; geriatric
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Letrozole; Anastrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): 90 days of pre-ET (endocrine therapy - tamoxifen or aromatase inhibitor) before Breast Cancer Surgery
  Interventions: Drug: Tamoxifen, Letrozole, Anastrozole, or Exemestane
- Control Arm (No Intervention): Will proceed directly to Breast Cancer Surgery

INTERVENTIONS:
Drug: Tamoxifen, Letrozole, Anastrozole, or Exemestane — Choice and dose of neoadjuvant endocrine therapy at the discretion of the treating medical oncologist.
  Other Names: Endocrine Therapy
  Arms: Intervention Arm

SUMMARY:
This is a Phase III, multisite exploratory study for women ≥ 65 years of age with early stage estrogen receptor positive (ER+) breast cancer. These individuals will be treated randomly assigned to one of two groups:

Intervention, treated with 3 months of pre-operative endocrine therapy (pre-ET) OR Control, participants follow standard of care and proceed directly to breast cancer surgery.

Both arms will be assessed for tolerance and compliance to the endocrine therapy by patient reported outcome (PRO) measures (patient surveys).

DETAILED DESCRIPTION:
Early-stage, estrogen receptor positive (ER+) breast cancer is traditionally treated with breast conserving surgery (BCS), radiation therapy (RT) and 5-10 years of adjuvant endocrine therapy (AET). Radiation therapy (RT) omission is an established treatment paradigm for women 65 years and older with ER+, node negative, small (≤ 3 cm) breast cancer. Despite the option for RT omission being recommended in the National Comprehensive Cancer Network (NCCN) guidelines, multiple modern studies demonstrate that a majority of older women still receive RT, raising concern for over-treatment. Conversely, there are a portion of patients who choose to omit RT but are not able to tolerate AET and thus are at risk for under-treatment and worse oncologic outcomes.

In the POWER I trial, patients were treated with 90 days of pre-operative endocrine therapy (pre-ET) as a window to establish endocrine therapy (ET) tolerance. The POWER I trial prospectively validated 90 days of pre-operative ET to determine if it could be used as a tool to inform adjuvant RT decisions and recommendations by patients and physicians respectively. Ninety days of pre-ET was shown to influence patient and physician preferences regarding adjuvant RT.

In the POWER II trial, participants will be randomized to treatment on either a) an intervention arm consisting of a 90-day window of pre-ET or b) the standard of care (control) arm in which participants proceed directly to BCS. In both arms, the decision to omit or administer adjuvant RT will be made by the treating physicians and patients. While not required per protocol, all patients will be recommended for AET if deemed appropriate by their oncologist, and adherence through 2 years will be monitored. The POWER I study revealed that pre-ET impacts patients' and physicians' decisions regarding adjuvant therapy and facilitates adjuvant therapy decisions that meld patient preferences and side effect tolerance. The purpose of the POWER II study is to examine whether 90 days of pre-ET results in a decrease in the number of (1) patients being treated with BCS alone and (2) patients treated with BCS+RT+AET. Adherence to AET will be defined as taking AET at 2 years post-BCS.

ELIGIBILITY:
Inclusion Criteria (summary):

* Diagnosis of ER+, PR +/-, and HER2- non amplified invasive breast cancer and clinically negative nodes
* ECOG performance status 0-2
* Females, aged ≥ 65 years
* Patient is eligible for BCS and opted for BCS
* Patient is a candidate for radiation therapy
* Patient is a candidate for endocrine therapy (tamoxifen or an aromatase inhibitor)
* Ability to take oral medication and be willing to adhere to endocrine therapy for the 3-month period prior to BCS
* Agreement to adhere to Lifestyle Considerations (details in protocol) throughout study duration
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Bilateral synchronous breast cancer
* Multicentric disease
* Prior use of SERMS or aromatase inhibitors
* History of ipsilateral breast radiation therapy
* Has a known additional malignancy that is progressing and/or requires active treatment with cytotoxic chemotherapy or radiation therapy. Malignancies deemed stable and low risk for complication per investigator's judgment may be allowed after discussion with multi-site PI.
* Current or planned use of a strong CYP2D6 inhibitor (e.g., Fluvoxamine, Paroxetine) and is not able to receive an endocrine therapy agent that does not use the CYP2D6 pathway.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2034-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who omit Radiation Therapy (RT) and are non-adherent to Endocrine Therapy (ET) | 24 months
  Proportion of participants who omit RT and are non-adherent to ET as measure through the 24-month adjuvant follow-up visit
Proportion of participants who are treated with Breast Cancer Surgery (BCS) + RT + AET | 24 months
  Proportion of participants who are treated with BCS + RT + AET as measured through the 24-month adjuvant follow-up visit

SECONDARY OUTCOMES:
Treatment with pre-ET and its impact on Decision Conflict | 24 months
  Using Patient Reported Outcomes (PRO) assessments of Decisional Conflict Scale (DCS) to determine whether treatment with pre-ET lessens Decision Conflict. The DCS is a validated measure of patient perceptions of uncertainty surrounding treatment choices. The minimum score is a 0, which is interpreted as no decisional conflict, and the maximum score is 64, which is interpreted as the highest decisional conflict.
Treatment with pre-ET and its impact on Decision Regret | 24 months
  Using Patient Reported Outcomes (PRO) assessments of Decision Regret Scale (DRS) to determine whether treatment with pre-ET lessens Decision Regret. The DRS is a validated, 5-item scale that measures self-reported regret after health care decisions. DRS scores range from 0 (no regret) to 100 (high regret).
Assessing whether patient's final treatment correlates with their beliefs about breast cancer | 7 months
  Using the PRO assessment "Beliefs about Illness Questionnaire (BIP-Q)" to determine patient's beliefs about breast cancer. The BIP-Q is a validated survey to assess cognitive and emotional perceptions of illness.
Assessing whether patient's final treatment correlates with their beliefs about breast cancer | 7 months
  Using the PRO assessment "Beliefs about Medicine Questionnaire (BMQ)" to determine patient's beliefs about breast cancer. The BMQ is a validated survey designed to capture patients' perceptions about medicines and medicine adherence.
Assessing whether patient's final treatment correlates with their beliefs about breast cancer | 7 months
  Using the PRO assessment "Perceived Sensitivity to Medicine (PSM)" to determine patient's beliefs about breast cancer. The PSM is a validated 5-question survey designed to capture patients' opinions regarding their sensitivity to medications.
Assessing whether treatment with pre-ET leads to improved Health Related Quality of Life compared to those treated with standard of care | 24 months
  Using PRO Assessments: EORTC Quality of Life questionnaires (QLQ-C30) to determine whether treatment with pre-ET leads to improved health-related quality of life compared to those treated with standard of care
Assessing whether early side effects of ET correlate with patient treatment group within study arms | 24 months
  Using the PRO Assessment "Breast Cancer Prevention Trial Symptom Checklist (BCPT-SCL)" to assess whether early side effects of ET correlate with patient treatment group within study arms
Assessing whether early side effects of ET correlate with patient treatment group within study arms | 24 months
  Using the PRO Assessment "Center for Epidemiologic Study Depression Scale Revised (CESD-R)" to assess whether early side effects of ET correlate with patient treatment group within study arms
To obtain data on local recurrence | 5 years
  Local recurrence as measured through the 5 year adjuvant follow-up period
To obtain data on regional recurrence | 5 years
  Regional recurrence as measured through the 5 year adjuvant follow-up period
To obtain data on contralateral breast cancer | 5 years
  Contralateral breast cancer as measured through the 5 year adjuvant follow-up period
To obtain data on distant metastases | 5 years
  Distant metastases as measured through the 5 year adjuvant follow-up period
To obtain data on disease free survival | 5 years
  Disease free survival (DFS) as measured through the 5 year adjuvant follow-up period
To obtain data on cancer specific survival | 5 years
  Cancer specific survival as measured through the 5 year adjuvant follow-up period
To obtain data on overall survival | 5 years
  Overall survival (OS) as measured through the 5 year adjuvant follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Shayna L Showalter, MD, Principal Investigator — University of Virginia
Locations (3):
- United States (3):
  - University of Virginia, Charlottesville, Virginia
  - INOVA Schar Cancer, Fairfax, Virginia
  - Virginia Commonwealth University, Richmond, Virginia